CLINICAL TRIAL: NCT04007029
Title: Study of CD19/CD20 Bispecific Chimeric Antigen Receptor (CAR)-T Cells for the Treatment of Relapsed or Refractory B-Cell Lymphomas and Chronic Lymphocytic Leukemia (CD20 - Cluster of Differentiation Antigen 20)
Brief Title: Modified Immune Cells (CD19/CD20 CAR-T Cells) in Treating Patients With Recurrent or Refractory B-Cell Lymphoma or Chronic Lymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Parker Institute for Cancer Immunotherapy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-001989; NCI-2019-03190 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18-001989 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2019-06-20; First posted 2019-07-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-05

CONDITIONS: CD19 Positive; CD20 Positive; Recurrent Chronic Lymphocytic Leukemia; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Primary Mediastinal (Thymic) Large B-Cell Cell Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Diffuse Large B-Cell Lymphoma; Refractory Follicular Lymphoma; Refractory Mantle Cell Lymphoma; Refractory Primary Mediastinal (Thymic) Large B-Cell Cell Lymphoma; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — Immunotherapy, Adoptive; Cyclophosphamide; fludarabine phosphate; tocilizumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (fludarabine, cyclophosphamide, CD19/CD20 T-cells) (Experimental): CONDITIONING CHEMOTHERAPY: Patients receive fludarabine phosphate IV over 30 minutes and cyclophosphamide IV over 60 minutes 5, 4, and 3 days before cell infusion.
  T-CELL INFUSION: Patients receive CD19/CD20 CAR-T cells IV on day 0. Patients with cytokine release syndrome may also receive tocilizumab IV on day 2 at the discretion of the clinical investigator.
  Interventions: Biological: Chimeric Antigen Receptor T-Cell Therapy; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Biological: Tocilizumab

INTERVENTIONS:
Biological: Chimeric Antigen Receptor T-Cell Therapy — Given Autologous anti-CD19/anti-CD20 CAR-expressing naive/memory T cells IV
  Other Names: CAR T Infusion; CAR T Therapy; CAR T-cell therapy; Chimeric Antigen Receptor T-cell Infusion
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP (cyclophosphamide) monohydrate; CTX (cytoxan); CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP fludarabine: 2-Fluoroadenine 9-beta-D-Arabinofuranoside 5'-Monophosphate; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Biological: Tocilizumab — Given IV
  Other Names: Actemra; Immunoglobulin G1, Anti-(Human Interleukin 6 Receptor) (Human-Mouse Monoclonal MRA Heavy Chain), Disulfide with Human-Mouse Monoclonal MRA Kappa-Chain, Dimer; MRA (myeloma receptor antibody); R-1569; RoActemra

SUMMARY:
This phase I trial studies the side effects and best dose of CD19/CD20 chimeric antigen receptor (CAR) T-cells when given together with chemotherapy, and to see how effective they are in treating patients with non-Hodgkin's B-cell lymphoma or chronic lymphocytic leukemia that has come back (recurrent) or has not responded to treatment (refractory). In CAR-T cell therapy, a patient's white blood cells (T cells) are changed in the laboratory to produce an engineered receptor that allows the T cell to recognize and respond to CD19 and CD20 proteins. CD19 and CD20 are commonly found on non-Hodgkin?s B-cell lymphoma and chronic lymphocytic leukemia cells. Chemotherapy drugs such as fludarabine phosphate and cyclophosphamide can control cancer cells by killing them, by preventing their growth, or by stopping them from spreading. Combining CD19/CD20 CAR-T cells and chemotherapy may help treat patients with recurrent or refractory B-cell lymphoma or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of the autologous anti-CD19/anti-CD20 CAR-expressing naive/memory T cells (CART19/20), including determination of the maximum tolerated dose and assessment for replication competent lentivirus (RCL).

SECONDARY OBJECTIVES:

I. Clinical response. Ia. Overall response rate. Ib. Duration of remission. Ic. Progression-free survival. Id. Overall survival. II. CD19/CD20 bispecific CAR transgenic T-cell persistence. IIa. T-cell monitoring and analyses. IIb. Evidence of B-cell aplasia.

EXPLORATORY OBJECTIVES:

I. To determine the serum levels of cytokines associated with cytokine release syndrome (CRS) in subjects exhibiting > grade-2 CRS following CART19/20 cell treatment.

OUTLINE: This is a dose-escalation study of CD19/CD20 CAR-T cells.

CONDITIONING CHEMOTHERAPY: Patients receive fludarabine phosphate intravenously (IV) over 30 minutes and cyclophosphamide IV over 60 minutes 5, 4, and 3 days before cell infusion.

T-CELL INFUSION: Patients receive CD19/CD20 CAR-T cells IV on day 0. Patients with cytokine release syndrome may also receive tocilizumab IV on day 2 at the discretion of the clinical investigator.

After completion of study treatment, patients are followed up daily for 14 days, on days 30, 45, 60, 70, 90, and 120, every 3 months for 2 years, every 6 months for 3 years, and then annually for a minimum of 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Diffuse large B-cell lymphoma (DLBCL), primary mediastinal large B-cell lymphoma (PMBCL), mantle cell lymphoma (MCL), follicular lymphoma (FL), chronic lymphocytic leukemia (CLL), or small lymphocytic lymphoma (SLL) that is refractory to standard-of-care options

  * DLBCL and PMBCL: primary refractory; relapsed after two prior lines of therapy
  * MCL, FL, CLL, and SLL: primary refractory; relapsed after three or more prior rounds of therapy
* > 30% positivity in malignant cells of either CD19 and/or CD20
* Minimum tumor burden of 1.5 cm^3 for lymphoma
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate bone marrow and major organ function to undergo a T cell transplant determined within 30?60 days prior to enrollment using standard phase I criteria for organ function. Blood may be evaluated while a patient is receiving growth factor support. Patients will be re-evaluated for organ function within 14 days of beginning conditioning chemotherapy
* Absolute neutrophil count (ANC) >= 1 x 10^9 cells/L (within 30-60 days prior to enrollment)
* Platelets >= 75 x 10^9/L (within 30-60 days prior to enrollment)
* Hemoglobin >= 8 g/dL (with or without transfusion) (within 30-60 days prior to enrollment)
* Aspartate and alanine aminotransferases (AST, ALT) =< 2.5 x upper limit of normal (ULN) (within 30-60 days prior to enrollment)
* Total bilirubin =< 2 x ULN (except patients with documented Gilbert?s syndrome) (within 30-60 days prior to enrollment)
* Creatinine < 2 mg/dL (or a glomerular filtration rate > 45) (within 30-60 days prior to enrollment)
* Must be willing and able to accept at least one leukapheresis procedure
* Must be willing and able to provide written informed consent

Exclusion Criteria:

* Inability to purify >= 1 x 10^7 T cells from leukapheresis product
* Previously known hypersensitivity to any of the agents used in this study; known sensitivity to cyclophosphamide or fludarabine
* Received systemic treatment for cancer, including immunotherapy, within 14 days prior to initiation of conditioning chemotherapy administration within this protocol. Patients who have received anti-CD19 CAR T-cells will be excluded from this trial. Consistent with current trials, patients may otherwise be given bridging therapy at the discretion of the lead study investigator
* Patients who have received an allograft transplant will NOT be allowed to participate in the trial. Patients who have received an autologous transplant will not be excluded and may participate in the trial
* Potential requirement for systemic corticosteroids or concurrent immunosuppressive drugs based on prior history or received systemic steroids within the last 2 weeks prior to enrollment (inhaled or topical steroids at standard doses are allowed)
* Human immunodeficiency virus (HIV) seropositivity or other congenital or acquired immune deficiency state, which would increase the risk of opportunistic infections and other complications during chemotherapy-induced lymphodepletion. If there is a positive result in the infectious disease testing that was not previously known, the patient will be referred to their primary physician and/or infectious disease specialist
* Hepatitis B or C seropositivity with evidence of ongoing liver damage, which would increase the likelihood of hepatic toxicities from the chemotherapy conditioning regimen and supportive treatments. If there is a positive result in the infectious disease testing that was not previously known, the patient will be referred to their primary physician and/or infectious disease specialist
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol
* Known clinically active brain metastases. Prior evidence of brain metastasis successfully treated with surgery or radiation therapy will not be exclusion for participation as long as they are deemed under control at the time of study enrollment and there are no neurological signs of potential brain metastases. A brain magnetic resonance imaging (MRI) scan taken within 60 days of screening may be used, otherwise a brain MRI must be performed to confirm absence of brain metastases
* A Tiffeneau-Pinelli index < 70% of the predicted value. Subjects will be excluded if pulmonary function tests indicate they have insufficient pulmonary capability
* A left ventricular ejection fraction as determined by an echocardiogram lower than 40% would preclude participation
* Pregnancy or breast-feeding. Female patients must be surgically sterile or be postmenopausal for two years, or must agree to use effective contraception during the period of treatment and for 6 months afterwards. All female patients with reproductive potential must have a negative pregnancy test (serum/urine) at screening and again within 14 days from starting the conditioning chemotherapy. The definition of effective contraception will be based on the judgment of the study investigators. Patients who are breastfeeding are not allowed on this study
* History of other malignancy in the past 3 years with the following exceptions:

  * Malignancy treated with curative intent and no known active disease
  * Adequately treated non-melanoma skin cancer without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
  * Adequately treated breast ductile carcinoma without evidence of disease
  * Prostate cancer with a Gleason score less than 6 with undetectable prostate specific antigen over 12 months
  * Adequately treated urothelial non-invasive carcinoma or carcinoma in situ
  * Similar neo-plastic conditions with an expectation of greater than 95% disease free survival

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-10-04 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 28 days from infusion
  Will be assessed according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, with the exception of cytokine release syndrome (CRS), which will be graded on the American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Grading for CRS scale. Simple descriptive statistics will be used to summarize toxicities observed after each transgenic T-cell infusion in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity (by CTCAE toxicity table) and minimum or maximum values for laboratory measures, time of onset, duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects. Adverse events will be tabulated by treatment group and will include the number of patients for whom the event occurred, the rate of occurrence, and the severity and relationship to study drug.
Dose-limiting toxicities | Up to 28 days from infusion
  Will be assessed per CTCAE version 5.0 with the exception of CRS as mentioned above.

SECONDARY OUTCOMES:
Clinical response | Up to 15 years
  Descriptive statistics including simple summary measures and plots appropriate for longitudinal data will be used.
Duration of remission | Time from complete remission (CR)/partial remission (PR) measurement criteria are first met until the first date that recurrent or progressive disease is objectively documented, or until death, assessed up to 15 years
  Descriptive statistics including simple summary measures and plots appropriate for longitudinal data will be used. Will also be summarized descriptively (mean, standard deviation, median, first and third quartiles, minimum, maximum). Figures showing the Kaplan-Meier estimates will also be presented.
Objective response rate (ORR) | Up to 15 years
  Descriptive statistics including simple summary measures and plots appropriate for longitudinal data will be used. ORR and the individual rate for CR and PR will be summarized with the frequency count and the percentage of subjects in each category, along with a 2-sided 95% exact confidence interval.
Progression-free survival | From time of study entry to documentation of objective disease progression or death due to any cause assessed up to 15 years
  Descriptive statistics including simple summary measures and plots appropriate for longitudinal data will be used. Will also be summarized descriptively (mean, standard deviation, median, first and third quartiles, minimum, maximum). Figures showing the Kaplan-Meier estimates will also be presented.
Overall survival (OS) | From date of enrollment until death, assessed up to 15 years
  Descriptive statistics including simple summary measures and plots appropriate for longitudinal data will be used. Will be summarized with figures using the Kaplan-Meier method. The Kaplan-Meier estimates for the 1-year OS (rates and the 2-sided 95% confidence interval of the rates using the Greenwood?s formula will be reported. Will also be summarized descriptively (mean, standard deviation, median, first and third quartiles, minimum, maximum).
Chimeric antigen receptor (CAR) T-cell (T) 19/20 bispecific transgenic T-cell persistence | Up to 5 years post-infusion
  Descriptive statistics of T-cell counts over time, including simple summary measures and plots appropriate for longitudinal data will be used.
Frequency of T cell phenotypic markers on CART19/20 cells using flow cytometry | Up to 5 years post-infusion
  The frequency of CART19/20 cell properties will be assessed using flow cytometry to indicate the % and/or total number of CART19/20 cells expressing critical markers, for example CD3 (cluster of differentiation 3), CD4 (cluster of differentiation 4), and CD8 (cluster of differentiation 8), to determine correlations between CART19/20 properties, treatment efficacy, and CART19/20 cell persistence.
Duration of B-cell aplasia following CART19/20 infusion. | Up to 2 years post-infusion
  The duration of time patients experience B-cell aplasia (<3% of lymphocytes in the peripheral blood expressing either CD19 or CD20, measured with immunohistochemistry (IHC) and/or flow cytometry) following infusion of CART19/20 cells will be determined.

OTHER OUTCOMES:
Analysis of proteins/cytokines (c-reactive protein (CRP), interleukin 6 (IL-6), tumor necrosis factor-alpha (TNF-α), and interferon-gamma (IFN-γ)) concentration in peripheral blood following CART19/20 infusion. | Up to 30 days post-infusion
  The cytokine levels in patients who receive CAR therapies will be monitored to help clarify the complex relationship between CRS severity, toxicity, T-cell survival, and disease eradication. Cytokine levels will be quantified in patients exhibiting any > grade-2 CRS. Cytokine levels in patients who do not exhibit CRS, or exhibit =< grade-2 CRS, will be quantified at the discretion of the investigator. The concentration in blood of each protein will be measured (CRP: mg/dL; IL-6, TNF-α, IFN-γ: pg/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Larson, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States